CLINICAL TRIAL: NCT06846931
Title: Comparison of the Efficacy of Low Intensity ESWT and Low Intensity LASER Therapy in the Treatment of Chronic Plantar Fasciitis; Randomized Controlled Trial
Brief Title: Comparison of the Efficacy of Shock Wave Therapy and Laser Therapy for Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Esat POLAT, Principal Investigator, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AhiEvranUERH-FTR-EP-01
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-02

CONDITIONS: Plantar Fasciitis, Chronic
Keywords: Rehabilitation; Extracorporeal Shock Wave Therapy; Low Intensity Laser; Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Extracorporeal Shockwave Therapy; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Three groups with a exercise control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Extracorporeal Shock Wave Therapy Group (Active Comparator): By the same physiotherapist with more than 5 years of clinical experience, radial ESWT treatment with 2500 pulses, 10 Hz frequency, 2.5-3 bar pressure, is applied to the most painful point of the heel and surrounding soft tissues, plantar aponeurosis and Achilles tendon insertion area on the dorsum of the heel, once a week for a total of 3 sessions. Plantar fascia stretching exercises (exercises to stretch the membrane on the sole of the foot), gastrocsoleus stretching exercises (exercises to stretch the calf muscles), foot intrinsic muscle strengthening exercises (exercises to strengthen the muscles on the sole of the foot) are taught to the patients by the doctor and they are asked to perform them 2 times a day 10 times for a total of 3 weeks.
  Interventions: Other: Extracorporeal Shock Wave Therapy; Other: EXERCİSE
- Low Intensity Laser Group (Active Comparator): A total of 28j (5.6jx5 points) are applied to the plantar fascia at 5 points on the heel by the same physiotherapist for 3 weeks, a total of 9 sessions (every other day) with the patient lying face down. Plantar fascia stretching exercises (exercises to stretch the membrane on the sole of the foot), gastrocsoleus stretching exercises (exercises to stretch the calf muscles), foot intrinsic muscle strengthening exercises (exercises to strengthen the muscles on the sole of the foot) are taught to the patients by the doctor and they are asked to perform them 2 times a day 10 times for a total of 3 weeks.
  Interventions: Other: Low Intensity Laser; Other: EXERCİSE
- Exercise Group (Placebo Comparator): Exercise therapy is carried out by the patient for 3 weeks. Plantar fascia stretching exercises (exercises to stretch the membrane on the sole of the foot), gastrocsoleus stretching exercises (exercises to stretch the calf muscles), foot intrinsic muscle strengthening exercises (exercises to strengthen the muscles on the sole of the foot) are taught to the patients by the doctor and they are asked to perform them 2 times a day 10 times for a total of 3 weeks.
  Interventions: Other: EXERCİSE

INTERVENTIONS:
Other: Extracorporeal Shock Wave Therapy — By the same physiotherapist with more than 5 years of clinical experience, radial ESWT treatment with 2500 pulses, 10 Hz frequency, 2.5-3 bar pressure, is applied to the most painful point of the heel and surrounding soft tissues, plantar aponeurosis and Achilles tendon insertion area on the dorsum of the heel, once a week for a total of 3 sessions.
  Arms: Extracorporeal Shock Wave Therapy Group
Other: Low Intensity Laser — A total of 28j (5.6jx5 points) are applied to the plantar fascia at 5 points on the heel by the same physiotherapist for 3 weeks, a total of 9 sessions (every other day) with the patient lying face down.
  Arms: Low Intensity Laser Group
Other: EXERCİSE — Exercise therapy is carried out by the patient for 3 weeks. Plantar fascia stretching exercises (exercises to stretch the membrane on the sole of the foot), gastrocsoleus stretching exercises (exercises to stretch the calf muscles), foot intrinsic muscle strengthening exercises (exercises to strengthen the muscles on the sole of the foot) are taught to the patients by the doctor and they are asked to perform them 2 times a day 10 times for a total of 3 weeks.

SUMMARY:
The aim of this study was to investigate the effects of extracorporeal shock wave therapy and low-intensity laser therapy on pain, functionality, plantar fascia thickness and balance in patients with plantar fasciitis.

DETAILED DESCRIPTION:
Plantar fasciitis is a pathology resulting from inflammation and/or degeneration of the plantar fascia of the sole of the foot. It affects about 10% of the population. It is one of the most common causes of chronic heel pain in the community and there is tenderness to palpation on the medial aspect of the heel bone. Patients complain of pain particularly with the first step in the morning and after rest. Mechanical overload and overuse can cause inflammation of the fascia. Diagnosis is usually made by clinical assessment and no further investigations are required.

In this study, 90 patients between the ages of 18 and 65 who meet the inclusion and exclusion criteria will be enrolled and participants will be randomised into 3 groups. The 1st group will be taught ESWT and home exercises for 1 session per week for 3 weeks and will be asked to do it every day. The 2nd group will receive 3 sessions of low intensity LASER per week for 3 weeks and will be asked to do home exercises every day. The 3rd group will only be taught home exercises and asked to do participants every day for 3 weeks. Visual analogue scale, foot function index, plantar fascia thickness measurement with USG and balance parameters will be measured at the beginning of the study, at the end of the treatment and at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 65 years of age, diagnosed with "plantar fasciitis" by anamnesis and physical examination
* Complaint duration of at least 3 months
* Patients who agree to participate in the study

Exclusion Criteria:

* Complaint lasting less than 3 months
* Injection in the heel area in the last 6 months
* Use of physiotherapy modalities for the heel in the last 6 months
* Bilateral complaint
* Pregnancy
* Malignancy
* Epilepsy
* History of cardiac pacemaker
* Anticoagulant use
* History of systemic inflammatory disease
* History of lower extremity fracture or surgery
* Existing open wound in the heel area
* Patient hypersensitivity
* Systemic infection in the patient
* Uncontrolled hypertension in the patient
* Patient inability to cooperate
* History of neuromuscular disease affecting balance parameters
* Unwillingness of the patient to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Before treatment (Week 0), at the end of treatment (Week 3) and after treatment (Week 12)
  On the VAS (Visual Analogue Scale), pain intensity is usually rated from 0 for "no pain" to 10 for "the worst pain imaginable" (10 cm scale). Scoring intervals for pain intensity: <3 mild pain, 3-6 moderate pain, >6 severe pain. The VAS is a practical scale that is widely used in chronic pain worldwide. In this study it is evaluated as Visual Analog Scale-rest (VAS-I), Visual Analog Scale-first press (VAS-ib) and Visual Analog Scale-activity (VAS-a).

SECONDARY OUTCOMES:
Foot Fonction Index | Before treatment (Week 0), at the end of treatment (Week 3) and after treatment (Week 12)
  It consists of 23 items with 3 subscales: pain, disability and activity limitation. The pain subscale, with nine items, measures the level of foot pain in different situations. The nine item disability subscale measures the degree of difficulty in performing various functional activities due to foot problems. The five-item Activity limitation subscale assesses activity limitations due to foot problems.
Plantar Fascia Thickness Measurement with Ultrasound Imaging | Before treatment (Week 0) and after treatment (Week 12)
  Ultrason görüntüleme PF tanısında, ayırıcı tanıda yumuşak doku patolojisinin dışlanmasında ve tedavinin takibinde kullanılabilir. Plantar fasya kalınlığının 4 mm'den fazla olması, Doppler modunda artmış kan akımı ve USG'de plantar fasyada hipoekoik alanlar PF tanısında önemlidir. Bu çalışmada, ayak bileği 90 derece dorsifleksiyonda iken yüzüstü pozisyonda longitudinal eksende kalınlık ölçülür. Fasya kalınlığı plantar fasyanın kalkaneal insersiyosunda ölçülecektir.
Measurement of Balance Parameters in Biodex Balance Device | Before treatment (Week 0), at the end of treatment (Week 3) and after treatment (Week 12)
  In a study conducted by Ağırman et al in 2019, plantar fasciitis was found to increase fall risk and negatively affect balance in the population under 65 years of age. In this study, postural stability and fall risk (total score, anteroposterior, mediolateral and overall stability) are assessed using the Bioedex balance device.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kirşehi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No